CLINICAL TRIAL: NCT02122276
Title: Effects of Continuous Passive Motion on the Spinal Circuitries and Its Adaptation in Patients With Spasticity Resulting From Upper Motor Neuron Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 96-1434B
Record Dates: First submitted 2014-04-17; First posted 2014-04-24 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Spinal Cord Injury(SCI)
Keywords: Spinal cord injury; Passive motion; Fatigue index; Hypertonia
MeSH Terms: conditions — Spinal Cord Injuries; Muscle Hypertonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SCI (Experimental): SCI participated in a 4-month robot-assisted passive ankle exercise regimen.
  Interventions: Procedure: Ankle continuous passive motion machine.

INTERVENTIONS:
Procedure: Ankle continuous passive motion machine. — A rehabilitation program of machine driven passive stretch exercise on ankle.

SUMMARY:
In animal and human studies, histochemical and physiological evidences showed that the muscle transferred from slow, fatigue-resistant muscle to fast, fatigable muscle after spinal cord injury. The alternation of muscular property was accompanied by the alternation of spinal circuitry property, and was related to the immobilization adaptation. Previous study showed that remobilization by continuous passive motion (CPM) for one month would restore the function of spinal circuitry in individual with chronic SCI. It is possible that long term application of CPM can reverse the adaptation of contractile properties of the paralyzed muscle after SCI. The purpose of this study is to investigate the effect of a four month CPM training on muscular properties in individuals with chronic SCI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of complete spinal cord injury

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The contractile properties of the muscles | Baseline, 1 month, 2 months, 3 months, and 4 months
  Measure of changes in contractile properties of soleus and tibialis anterior
Fatigue index | Baseline, 1 month, 2 months, 3 months, and 4 months
  Measure of changes in Fatigue index of soleus and tibialis anterior.
Clinical muscle tone tests | Baseline, 1 month, 2 months, 3 months, and 4 months
  Measure of changes in clinical muscle tone tests of soleus and tibialis anterior by Modified Ashworth Scale.
Patient Reported Impact of Spasticity Measure (PRISM) | Baseline, 1 month, 2 months, 3 months, and 4 months
  Measure of changes in PRISM.
The potential adverse effects of ankle swelling | Baseline, 1 month, 2 months, 3 months, and 4 months
  Measure of changes in the potential adverse effects of ankle swelling.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan